CLINICAL TRIAL: NCT06605391
Title: Caregiving While Black-LIVE: Empowering Black Dementia Caregivers to Navigate Care
Brief Title: Caregiving While Black: LIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Fayron Epps, Adjunct Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005946; R21AG083366 (NIH)
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Results first posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Dementia
Keywords: Caregiving
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregiving While Black-LIVE (Experimental): Black dementia caregivers participating in the psychoeducation course, Caregiving while Black-LIVE, over an 8 week time period.
  Interventions: Behavioral: Caregiving While Black-LIVE

INTERVENTIONS:
Behavioral: Caregiving While Black-LIVE — Caregiving while Black-LIVE is a psychoeducation program that aims to intensify the development of caregiver mastery by integrating the online learning assets of the fully asynchronous Caregiving while Black program with synchronous, group-based opportunities for interactivity and active learning. The Caregiving while Black course includes topics of navigating the healthcare system, managing home life, and caregiver self-care. Once enrolled in the course, participants will be provided instructions for accessing the weekly sessions and course online, and supplemental course materials will be mailed to them. The Canvas platform enables the research team to monitor each individual's movement in the cohort through the asynchronous part of the course. Nudges and reminders to view these materials are sent twice a week via text or email with participant's consent. Synchronous sessions are conducted on a videoconferencing platform.

SUMMARY:
This study will test the psychoeducation course, Caregiving while Black - Learning In Vital Engagement (LIVE), among Black caregivers providing care to persons with dementia. This course aims to enhance Black caregivers' capacity to cope effectively with their caregiving role of navigating care and the world of healthcare in ways that take into consideration the social and cultural context of their unique life experiences.

DETAILED DESCRIPTION:
Black caregivers and their care recipients experience disparities in care, have lower rates of formal service use, and are generally under-treated. More specifically, disparities in healthcare quality include higher rates of missed or delayed dementia diagnoses among Black older adults and a lower likelihood of receiving dementia medication or care from a dementia specialist. Notably, disparities exist for caregivers of persons living with Alzheimer's disease and persons living with dementia (PLWD) as well: Black caregivers report more time spent in caregiving than do White caregivers and use less respite service. Black caregivers also report increased difficulties navigating the healthcare system. Further, racial differences and disparities related to caregiving experiences exist at alarming rates for use of supportive services (33% vs 25%), care hours (54% vs 39%), and living below the federal poverty level (32% vs 12%) among Black caregivers compared to White caregivers. Black families faced with dementia (Medicare beneficiaries) incur 1.7 times more in healthcare cost and higher proportions of preventable hospitalizations than White families. Among PLWD, Black older adults account for nearly a third of preventable hospitalizations. It should be noted that these disparities are not due to biological or genetic differences between racial or ethnic groups, as race and ethnicity are social constructs. Rather, it is more likely due to lived experience and structural racism leading to disparities in social and structural determinants of health. These amplified experiences highlight the importance of this proposal to further develop a course that addresses the cultural and practical reality of supporting a PLWD as a Black in America, as Black caregivers desire better access to culturally relevant caregiving and self-care information. One potential tool to mitigate the aforementioned health disparities is to offer an education tailored and responsive to the needs of Black caregivers. This project responds to a compound gap in psychoeducation aimed at promoting caregiving mastery.

This study will test the psychoeducation course, Caregiving while Black - LIVE, among Black caregivers providing care to persons with dementia. The researchers will employ a mixed-methods pre-post no control design to gather formative and evaluative data from four cohorts (10 participants in each cohort) of Black caregivers. The course is self-paced and participants are asked to complete the course over an 8-week period.

ELIGIBILITY:
Caregiver Inclusion Criteria:

* at least 18 years of age
* family member (or friend) who self-identifies as Black American and as the principal caregiver of a community-dwelling PLWD (not in hospice care) and who is the principal companion of that person during healthcare encounters
* provides some hands-on care multiple times a week
* has access to an electronic device and/or access to broadband internet
* able to speak and understand English

Caregiver Exclusion Criteria:

* persons who cannot provide consent

  * persons who are not yet adults (under 18 years of age)
  * prisoners
  * cognitively impaired adults
* have plans to relinquish caring responsibilities for PLWD or are considering moving the PLWD to an institutional setting within the next 6 months
* not able to clearly understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fayron Epps, PhD, RN, Principal Investigator — Emory University
Locations (1):
- Emory University, Nell Hodgson Woodruff School of Nursing, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be made available for sharing, after deidentification.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing beginning 3 months and ending 5 years following publication of findings from this study in a scientific journal.
Access Criteria: Data will be available for sharing with researchers who provide a methodologically sound proposal, for the purposes of achieving the aims in the approved proposal. Proposals should be directed to fepps@emory.edu. To gain access, data requestors will need to sign a data access agreement. Data will be available for 5 years at a third party website.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled through Emory University in Atlanta, Georgia, USA. Participant enrollment began October 1, 2024 and all follow-up assessments were completed by August 12, 2025.
Period: Overall Study
Arm/Group | Caregiving While Black-LIVE
Started | 40
Completed the Assessment at Month 3 | 36
Completed (Completed the assessment at Month 6) | 30
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.60 (9.75)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 34
  Male | 5
  Non-binary | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 40
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Relation to person living with dementia who is being cared for [Count of Participants; unit: Participants]
  Spouse | 5
  Parent | 29
  Other relative | 6
Living with person living with dementia [Count of Participants; unit: Participants]
  No | 21
  Yes | 19
Employed outside of the home [Count of Participants; unit: Participants]
  No | 15
  Yes | 25
Education [Count of Participants; unit: Participants]
  High school/General Educational Development (GED) | 1
  Some college | 8
  College graduate | 22
  Graduate degree | 9
Marriage status [Count of Participants; unit: Participants]
  Single | 13
  Married | 20
  Divorced or separated | 4
  Widowed | 3
Annual income [Count of Participants; unit: Participants]
  $0 - $30,000 | 7
  $31,000 - $60,000 | 10
  $61,000 - $90,000 | 6
  $91,000 - $120,000 | 9
  More than $120,000 | 4
  Do not wish to answer | 4
Area of residence [Count of Participants; unit: Participants]
  Urban | 14
  Suburban | 22
  Rural | 4

OUTCOME MEASURES:

1. Primary Outcome: Health Literacy Questionnaire (HLQ) Score for Feeling Understood by Healthcare Providers Subscale
Description: The Health Literacy Questionnaire assesses multiple dimensions of health literacy with 9 subscales. The subscale of "Feeling understood and supported by healthcare providers" has 4 items where responses are given on a 4-point scale from "strongly disagree" (scored as 1) to "strongly agree" (scored as 4). The total score for this subscale is the average of responses and ranges from 1 to 4. Higher scores indicate that the subscale is an area of health literacy strength.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
score on a scale
  Baseline | 3.0 (0.71)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 2.9 (0.69)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 3.0 (0.61)

2. Primary Outcome: Health Literacy Questionnaire (HLQ) Score for Appraisal of Health Information Subscale
Description: The Health Literacy Questionnaire assesses multiple dimensions of health literacy with 9 subscales. The subscale of "Appraisal of health information" has 5 items where responses are given on a 4-point scale from "strongly disagree" (scored as 1) to "strongly agree" (scored as 4). The total score for this subscale is the average of responses and ranges from 1 to 4. Higher scores indicate that the subscale is an area of health literacy strength.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
score on a scale
  Baseline | 3.1 (0.61)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 3.2 (0.55)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 3.1 (0.37)

3. Primary Outcome: Health Literacy Questionnaire (HLQ) Score for Ability to Engage With Healthcare Providers Subscale
Description: The Health Literacy Questionnaire assesses multiple dimensions of health literacy with 9 subscales. The subscale of "Ability to actively engage with healthcare providers" has 5 items where responses are given on a 5-point scale from "cannot do" (scored as 1) to "very easy" (scored as 5). The total score for this subscale is the average of responses and ranges from 1 to 5. Higher scores indicate that the subscale is an area of health literacy strength.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
score on a scale
  Baseline | 3.9 (0.62)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 4.0 (0.64)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 4.1 (0.51)

4. Primary Outcome: Health Literacy Questionnaire (HLQ) Score for Navigating the Healthcare System Subscale
Description: The Health Literacy Questionnaire assesses multiple dimensions of health literacy with 9 subscales. The subscale of "Navigating the healthcare system" has 6 items where responses are given on a 5-point scale from "cannot do" (scored as 1) to "very easy" (scored as 5). The total score for this subscale is the average of responses and ranges from 1 to 5. Higher scores indicate that the subscale is an area of health literacy strength.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
score on a scale
  Baseline | 3.5 (0.62)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 3.7 (0.51)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 3.7 (0.49)

5. Primary Outcome: Health Literacy Questionnaire (HLQ) Score for Ability to Find Information Subscale
Description: The Health Literacy Questionnaire assesses multiple dimensions of health literacy with 9 subscales. The subscale of "Ability to find good health information" has 5 items where responses are given on a 5-point scale from "cannot do" (scored as 1) to "very easy" (scored as 5). The total score for this subscale is the average of responses and ranges from 1 to 5. Higher scores indicate that the subscale is an area of health literacy strength.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
score on a scale
  Baseline | 3.8 (0.57)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 3.8 (0.39)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 4.0 (0.47)

6. Primary Outcome: Health Literacy Questionnaire (HLQ) Score for Understand Health Information Subscale
Description: The Health Literacy Questionnaire assesses multiple dimensions of health literacy with 9 subscales. The subscale of "Understand health information well enough to know what to do" has 5 items where responses are given on a 5-point scale from "cannot do" (scored as 1) to "very easy" (scored as 5). The total score for this subscale is the average of responses and ranges from 1 to 5. Higher scores indicate that the subscale is an area of health literacy strength.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
score on a scale
  Baseline | 4.0 (0.50)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 4.0 (0.41)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 4.1 (0.52)

7. Primary Outcome: Zarit Burden Inventory (ZBI) Score
Description: The Zarit Burden Interview is a 22-item scale of objective and subjective caregiver burden. Responses are given on a 5-point scale where 0 = never and 4 = nearly always. Total scores range from 0 to 88 where higher scores indicate greater feelings of being burdened with providing care.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
score on a scale
  Baseline | 34.2 (15.44)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 31.0 (11.95)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 29.8 (11.03)

8. Primary Outcome: Center for Epidemiological Studies - Depression Score
Description: Caregiver depression will be assessed with the 20-item Center for Epidemiologic Studies - Depression Scale. Caregivers are asked how frequently they have experienced specific symptoms of depression in the past week. Responses are given as 0 = rarely, 1 = 1-2 days, 2 = 3-4 days, and 4 = 5-7 days. Total scores range from 0 to 60 with higher scores indicating greater symptoms of depression.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
score on a scale
  Baseline | 11.8 (8.94)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 10.8 (8.39)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 8.6 (7.78)

9. Primary Outcome: Perceived Stress Scale Score
Description: Caregiver stress was assessed with the 14-item Perceived Stress Scale. Responses are given on a scale of 0 to 4 where 0 = never and 4 = very often. Total scores range from 0 to 56 with higher scores indicating greater perceived stress by caregivers.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
score on a scale
  Baseline | 24.8 (8.18)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 23.0 (7.35)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 22.6 (6.05)

10. Primary Outcome: State-Trait Anxiety Inventory (STAI) Score
Description: The STAI is a 20-item self-report scale of positive and negative anxiety experiences. Responses are given on a 4-point scale where 1 = not at all and 4 = very much so. Total scores range from 20 to 80 and higher scores indicate greater anxiety.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points. Two participants did not complete this assessment at the Baseline visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 38
score on a scale
  Baseline | 39.2 (12.30)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 36.2 (8.70)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 35.8 (7.92)

11. Primary Outcome: Caregiver Assessment of Behavioral Skill Score
Description: The Caregiver Assessment of Behavioral Skill instrument includes 17 items asking how frequently caregivers respond to certain situations. Responses are given on a 3-point scale where "seldom true" is scored as 0 and "true most of the time" is scored as 2 (a response is also available when the situation is not relevant). The total score is is the sum of item ratings and ranges from 0 to 34, where higher scores indicate greater behavioral skills as related to caregiving.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
score on a scale
  Baseline | 14.3 (5.33)
  Month 3: number analyzed (Participants) | 36
  Month 3 | 14.4 (4.57)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 14.9 (5.97)

12. Primary Outcome: Pearlin Competence and Management of Situation Score
Description: Self-rated caregiving competency is assessed with 4 items asking about feelings the caregiver has as a result of providing care. Responses are given on a 4-point scale where "not at all" is scored as 1 and "completely" or "very" is scored as 4. The total score ranges from 4 to 16 with higher scores indicating greater feelings of competency.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants who completed study assessment at the indicated time points. One participant did not complete this assessment at the Month 3 time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiving While Black-LIVE
Number analyzed (Participants) | 40
score on a scale
  Baseline | 11.8 (2.40)
  Month 3: number analyzed (Participants) | 35
  Month 3 | 13.4 (2.03)
  Month 6: number analyzed (Participants) | 30
  Month 6 | 13.5 (2.05)

13. Other Pre Specified Outcome: Change in Health Literacy Questionnaire (HLQ) Score for Social Support Subscale
Description: The Health Literacy Questionnaire assesses multiple dimensions of health literacy with 9 subscales. The subscale of "Social support for health" has 5 items where responses are given on a 4-point scale from "strongly disagree" (scored as 1) to "strongly agree" (scored as 4). The total score for this subscale is the average of responses. Higher scores indicate that the subscale is an area of health literacy strength.
Time Frame: Baseline, Month 3, Month 6
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Health Literacy Questionnaire (HLQ) Score for Actively Managing Health Subscale
Description: The Health Literacy Questionnaire assesses multiple dimensions of health literacy with 9 subscales. The subscale of "Actively managing my health" has 5 items where responses are given on a 4-point scale from "strongly disagree" (scored as 1) to "strongly agree" (scored as 4). The total score for this subscale is the average of responses. Higher scores indicate that the subscale is an area of health literacy strength.
Time Frame: Baseline, Month 3, Month 6
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Health Literacy Questionnaire (HLQ) Score for Having Sufficient Information Subscale
Description: The Health Literacy Questionnaire assesses multiple dimensions of health literacy with 9 subscales. The subscale of "Having sufficient information to manage my health" has 4 items where responses are given on a 4-point scale from "strongly disagree" (scored as 1) to "strongly agree" (scored as 4). The total score for this subscale is the average of responses. Higher scores indicate that the subscale is an area of health literacy strength.
Time Frame: Baseline, Month 3, Month 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information about adverse events was collected beginning at the Baseline assessment and ending at the Month 6 assessment, for a total of 6 months.
Arm/Group | Caregiving While Black-LIVE
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT06605391/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT06605391/ICF_000.pdf